CLINICAL TRIAL: NCT03944772
Title: A Biomarker-directed Phase 2 Platform Study in Patients With Advanced Non-Small Lung Cancer Whose Disease Has Progressed on First-Line Osimertinib Therapy.
Brief Title: Phase 2 Platform Study in Patients With Advanced Non-Small Lung Cancer Who Progressed on First-Line Osimertinib Therapy (ORCHARD)
Acronym: ORCHARD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6186C00001; 2023-504624-25-00 (Registry Identifier: CTIS); 2018-003974-29 (EudraCT Number)
Record Dates: First submitted 2019-04-29; First posted 2019-05-10 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-12

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-small cell lung cancer; NSCLC; tSCLC; NEC; Phase II; Platform study; Biomarker-directed; Durvalumab; Osimertinib; Savolitinib; Selumetinib; Etoposide; Gefitinib; Necitumumab; Platinum-containing doublet; Pemetrexed; EGFR positive; Carboplatin; Alectinib; Selpercatinib; Cisplatin; TKI-resistant; MET amplification; MET exon 14 skipping; EGFR; EGFR C797X; EGFR G724X; EGFR L718X; EGFR exon 20 insertion; EGFR amplification; BRAF V600E; ALK rearrangement; RET rearrangement; ROS1 rearrangement; NTRK fusion; KRAS G12C; Datopotamab deruxtecan
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib; 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine; Gefitinib; necitumumab; durvalumab; Carboplatin; Pemetrexed; alectinib; selpercatinib; AZD 6244; Etoposide; Cisplatin

STUDY DESIGN:
Intervention Model Description: Phase 2 platform study in patients with advanced Non-Small Lung Cancer harbouring an epidermal growth factor receptor (EGFR)-sensitizing mutation with evidence of radiological progression following first-Line osimertinib therapy. This study is modular in design, allowing evaluation of the efficacy, safety and tolerability of multiple study treatments. The study will be conducted in three groups (Groups A, B and C). Patient allocation to a study treatment within each group will be based on tumour molecular profile. Biomarker positive patients or patients with histologically identifiable neuroendocrine transformation to small cell lung cancer (SCLC) or large cell neuroendocrine carcinoma (NEC) will be allocated to a biomarker-matched study treatment in Group A, patients without a biomarker will be allocated to a study treatment in Group B and patients with a biomarker amenable to therapies not currently available in ORCHARD will be allocated to Group C.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Module 1: Osimertinib + Savolitinib (Experimental): The patients in this group will receive osimertinib taken in combination with savolitinib
  Interventions: Drug: Osimertinib; Drug: Savolitinib
- Module 2: Osimertinib + Gefitinib (Experimental): The patients in this group will receive osimertinib taken in combination with gefitinib
  Interventions: Drug: Osimertinib; Drug: Gefitinib
- Module 3: Osimertinib + Necitumumab (Experimental): The patients in this group will receive osimertinib taken in combination with necitumumab
  Interventions: Drug: Osimertinib; Drug: Necitumumab
- Module 4: Carboplatin + Pemetrexed + Durvalumab) (Experimental): The patients in this group will receive platinum-containing doublet (carboplatin + pemetrexed) taken in combination with durvalumab.
  Interventions: Drug: Durvalumab; Drug: Carboplatin; Drug: Pemetrexed
- Observational Cohort: No study drug (No Intervention): Patients in this group will not receive study treatment but receive further anticancer care (Standard of Care therapy or other experimental therapies) or supportive care, as clinically indicated, in accordance with local practice.
  With Group C, the aim is to understand the clinical course and/or outcome for the overall clinical population after progression on first-line monotherapy with osimertinib.
- Module 5: Osimertinib + Alectinib (Experimental): The patients in this group will receive osimertinib taken in combination with alectinib
  Interventions: Drug: Osimertinib; Drug: Alectinib
- Module 6: Osimertinib + Selpercatinib (Experimental): The patients in this group will receive osimertinib taken in combination with selpercatinib
  Interventions: Drug: Osimertinib; Drug: Selpercatinib
- Module 7: Etoposide + Durvalumab + Carboplatin or Cisplatin (Experimental): The patients in this group will receive platinum-containing doublet (etoposide + carboplatin or cisplatin) taken in combination with durvalumab.
  Interventions: Drug: Durvalumab; Drug: Carboplatin; Drug: Etoposide; Drug: Cisplatin
- Module 8: Osimertinib + Pemetrexed + Carboplatin or Cisplatin. (Experimental): The patients in this group will receive Osimertinib plus platinum-containing doublet (pemetrexed + carboplatin or cisplatin).
  Interventions: Drug: Osimertinib; Drug: Carboplatin; Drug: Pemetrexed; Drug: Cisplatin
- Module 9: Osimertinib + Selumetinib (Experimental): The patients in this group will receive osimertinib taken in combination with selumetinib
  Interventions: Drug: Osimertinib; Drug: Selumetinib
- Module 10: Osimertinib + datopotamab deruxtecan (Experimental): The patients in this group will receive osimertinib taken in combination with datopotamab deruxtecan.
  Interventions: Drug: Osimertinib; Drug: Datopotamab deruxtecan

INTERVENTIONS:
Drug: Osimertinib — Osimertinib given orally at 80 mg once daily
  Other Names: TAGRISSO
  Arms: Module 10: Osimertinib + datopotamab deruxtecan; Module 1: Osimertinib + Savolitinib; Module 2: Osimertinib + Gefitinib; Module 3: Osimertinib + Necitumumab; Module 5: Osimertinib + Alectinib; Module 6: Osimertinib + Selpercatinib; Module 8: Osimertinib + Pemetrexed + Carboplatin or Cisplatin.; Module 9: Osimertinib + Selumetinib
Drug: Savolitinib — Savolitinib will be given orally at 300 mg or 600mg once daily
  Arms: Module 1: Osimertinib + Savolitinib
Drug: Gefitinib — Gefitinib given orally at 250 mg once daily
  Other Names: Iressa
  Arms: Module 2: Osimertinib + Gefitinib
Drug: Necitumumab — Necitumumab given IV at 800 mg on Day 1 and Day 8 of every 3-week cycle
  Other Names: Portrazza
  Arms: Module 3: Osimertinib + Necitumumab
Drug: Durvalumab — Durvalumab given IV at 1500 mg on Day 1 of every cycle
  Other Names: IMFINZI
  Arms: Module 4: Carboplatin + Pemetrexed + Durvalumab); Module 7: Etoposide + Durvalumab + Carboplatin or Cisplatin
Drug: Carboplatin — Carboplatin given IV on Day 1 of every 21-day cycle for up to 6 cycles
  Arms: Module 4: Carboplatin + Pemetrexed + Durvalumab); Module 7: Etoposide + Durvalumab + Carboplatin or Cisplatin; Module 8: Osimertinib + Pemetrexed + Carboplatin or Cisplatin.
Drug: Pemetrexed — Pemetrexed given IV at 500 mg/m2 body BSA on Day 1 of every cycle
  Arms: Module 4: Carboplatin + Pemetrexed + Durvalumab); Module 8: Osimertinib + Pemetrexed + Carboplatin or Cisplatin.
Drug: Alectinib — Alectinib given orally at 600mg twice daily and for Japanese patients at 300mg twice daily.
  Other Names: Alecensa
  Arms: Module 5: Osimertinib + Alectinib
Drug: Selpercatinib — Selpercatinib given orally at 160mg twice daily
  Other Names: Loxo-292, Retevmo, Retsevmo
  Arms: Module 6: Osimertinib + Selpercatinib
Drug: Selumetinib — Selumetinib given orally at 75 mg twice daily for 4 days, followed by 3 days off treatment
  Other Names: Koselugo
  Arms: Module 9: Osimertinib + Selumetinib
Drug: Etoposide — Etoposide 80-100 mg/m2 given IV on day 1, 2 and 3 of every 21-day cycle for up to 4 cycles.
  Arms: Module 7: Etoposide + Durvalumab + Carboplatin or Cisplatin
Drug: Cisplatin — Cisplatin 75-80 mg/m2 given IV on days 1 of each cycle
  Arms: Module 7: Etoposide + Durvalumab + Carboplatin or Cisplatin; Module 8: Osimertinib + Pemetrexed + Carboplatin or Cisplatin.
Drug: Datopotamab deruxtecan — Datopotamab deruxtecan given IV at 4 or 6 mg/kg on Day 1 of every 3-week cycle.
  Other Names: DS 1062a
  Arms: Module 10: Osimertinib + datopotamab deruxtecan

SUMMARY:
Phase 2 Platform Study in Patients with Advanced Non-Small Lung Cancer who progressed on First-Line Osimertinib Therapy. This study is modular in design, allowing evaluation of the efficacy, safety and tolerability of multiple study treatments.

DETAILED DESCRIPTION:
This is an open-label, multicentre, multi-drug, biomarker-directed Phase 2 platform study in patients with advanced non-small cell lung cancer (NSCLC) harbouring an epidermal growth factor receptor (EGFR)-sensitizing mutation whose disease has progressed on first-line monotherapy with osimertinib.Treatment options for these patients are limited. Novel treatments for these patients are urgently required.

This study is modular in design, allowing evaluation of the efficacy, safety and tolerability of multiple study treatments.

ELIGIBILITY:
Inclusion criteria applicable to all study treatment modules (Group A & B)

1. NSCLC with the following features:

   1. Locally advanced or metastatic disease (ie, advanced NSCLC) not amenable to curative surgery or radiotherapy at study entry.
   2. Histologically or cytologically confirmed adenocarcinoma of the lung (patients with mixed histology are eligible if adenocarcinoma is the predominant histology) harboring EGFR mutation(s) known to be associated with EGFR TKI sensitivity at diagnosis. Any histologically identifiable component of neuroendocrine transformation to SCLC or large cell NEC is required for treatment under Module 7.
   3. Received only one line of therapy, with single-agent osimertinib, for advanced NSCLC, with clinical benefit as judged by investigator discretion.

      (Note: a 'line' of therapy is defined as a daily anti-cancer treatment administered for >14 days, or a single infusion of an intravenous anti-cancer treatment. For instance, patients who have had <14 days of a first- or second- generation TKI prior to osimertinib, and stopped due to adverse events, would be eligible to enter this study, see also exclusion criteria 5).

      Patients previously treated adjuvantly or neo-adjuvantly are eligible per exclusion criterion 5.
   4. Evidence of radiological disease progression on first-line monotherapy with osimertinib 80 mg po QD.
2. Suitable for a mandatory biopsy defined as having an accessible tumor; by whichever modality the site uses and, ideally, confirmed by the person who will perform the procedure; and a stable clinical condition that will allow the patient to tolerate the procedure. The biopsy should be performed within 60 days of the planned first dose of study treatment.
3. Patients must have measurable disease per RECIST 1.1, as defined by at least 1 lesion that can be accurately measured at baseline as ≥ 10 mm at the longest diameter (except lymph nodes which must have a short axis ≥ 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI), which is suitable for accurate repeated measurements. Previously irradiated lesions or a lesion in the field of radiation should not be used as measurable disease unless the lesion(s) has/have demonstrated unequivocal disease progression by RECIST 1.1. Target lesions should not be used for the baseline tumour biopsy, unless there are no other lesions suitable for biopsy and they fulfil requirements.
4. Adequate coagulation parameters, defined as:

International Normalisation Ratio (INR) < 1.5 × upper limit of normal (ULN) and activated partial thromboplastin time < 1.5 × ULN unless patients are receiving therapeutic anti-coagulation which affects these parameters.

-------------------------------------------------------------------------------------------

Exclusion Criteria applicable to all study treatment modules (Groups A/B):

1. Patients whose disease has progressed within the first 3 months of osimertinib treatment (refractory to osimertinib treatment).
2. Patients must not have experienced a toxicity(-ies) that led to permanent discontinuation or dose reduction of prior osimertinib.

   (a) Patients who had dose reductions in the past, but were receiving a full dose of osimertinib at the time of pre-screening should be discussed with the Study Physician.
3. Any unresolved toxicities from prior osimertinib treatment greater than CTCAE Grade 1 at the time of starting study treatment.
4. Patients should not have discontinued osimertinib >60 days prior to the first dose of study treatment.
5. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

   1. Absolute neutrophil count < 1.5 × 109/L.
   2. Platelet count < 100 × 109/L.
   3. Haemoglobin < 9 g/dL.
   4. Alanine transaminase (ALT) > 2.5 × ULN.
   5. Aspartate aminotransferase (AST) > 2.5 × ULN.
   6. Total bilirubin (TBL) > 1.5 × ULN, or > 3 × ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinaemia).
6. Creatinine clearance (CrCl) < 50 mL/min, calculated using Cockcroft-Gault equation (Cockcroft and Gault 1976) or 24-hour urine collection. For medical conditions where the Cockcroft-Gault equation is inappropriate or 24-hour urine collection is unfeasible, CrCl may be calculated differently following written approval from the Study Physician.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2025-05-06 (Estimated); Study Completion 2025-05-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Measured from first dose until confirmed response or progression. For each patient this is expected to be 3 months on average
  The percentage of patients with a confirmed investigator-assessed complete or partial response according to Response Evaluation Criteria In Solid Tumours (RECIST) 1.1. Patients will be followed up every 6 weeks (±1 week) for the first 24 weeks and every 9 weeks thereafter until RECIST 1.1 defined disease progression or cessation of study treatment (if treating beyond progression).

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Measured from first dose until progression. For each patient this is expected to be 6 months on average
  The time from first dose until the date of objective disease progression or death (by any cause in the absence of progression). Patients will be followed up every 6 weeks (±1 week) for the first 24 weeks and every 9 weeks thereafter until RECIST (Response Evaluation Criteria In Solid Tumours)1.1 defined disease progression or cessation of study treatment (if treating beyond progression).
Duration of response (DoR) | Measured from response until progression. For each patient this is expected to be 6 months on average
  The time from the date of first response until date of disease progression or death in the absence of disease progression. Patients will be followed up every 6 weeks (±1 week) for the first 24 weeks and every 9 weeks thereafter until RECIST 1.1 defined disease progression or cessation of study treatment (if treating beyond progression).
Overall survival (OS) | Measured from first dose until death or final cohort data cut-off. For each patient this is expected to be 20 months on average
  The time from the date of the first dose of study treatment until death due to any cause.
Plasma/serum concentrations of therapeutic agents | Pre-dose and 1 hour post-dose blood samples on Day 1 of Cycles 1, 3 (Cycle 2 for durvalumab), 6 for all therapeutic agents and a sample at the 90-day safety follow up for durvalumab only. (One Cycle = 21 or 28 days, depending on treatment).
  Blood samples will be collected at various timepoints to evaluate the sparse pharmacokinetics of study therapeutic agents.
Plasma/serum concentrations of therapeutic agents | Pre-dose and serial post-dose blood samples (1 hour, 2 hours, 4 hours, 6 hours, 8 hours) on Day 15 of Cycle 1 for alectinib and selpercatinib only.
  Blood samples will be collected at various timepoints to evaluate the serial pharmacokinetics of study therapeutic agents
Incidence of Treatment-emergent adverse events (AEs) and serious adverse events (SAEs) as characterized and graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Event [CTCAE] v5 | Continuously from first dose to end of safety follow up after study treatment discontinuation (approximately up to 21 Months)
  To evaluate safety and tolerability of each study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Helena A Yu, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center, 1275 York Avenue, New York, NY 10065, USA
Locations (40):
- United States (14):
  - Research Site, Duarte, California
  - Research Site, Los Angeles, California
  - Research Site, Sacramento, California
  - Research Site, Santa Monica, California
  - Research Site, New Haven, Connecticut
  - Research Site, Chicago, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Grand Rapids, Michigan
  - Research Site, New York, New York
  - Research Site, Portland, Oregon
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Houston, Texas
  - Research Site, Seattle, Washington
- Research Site, Odense C, Denmark
- Italy (5):
  - Research Site, Catania
  - Research Site, Napoli
  - Research Site, Orbassano
  - Research Site, Padua
  - Research Site, Varese
- Japan (6):
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Kōtoku
  - Research Site, Nagoya
  - Research Site, Osaka
  - Research Site, Wakayama
- Netherlands (4):
  - Research Site, Amsterdam
  - Research Site, Maastricht
  - Research Site, Nijmegen
  - Research Site, Rotterdam
- Norway (3):
  - Research Site, Drammen
  - Research Site, Oslo
  - Research Site, Trondheim
- South Korea (2):
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (4):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Seville
- Research Site, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Riess JW, de Langen AJ, Ponce S, Goldberg SB, Piotrowska Z, Goldman JW, Le X, Cho BC, Yoneshima Y, Ambrose H, Cavazzina R, Tang KH, Lau J, Yu HA. ORCHARD: Osimertinib Plus Necitumumab in Patients With Epidermal Growth Factor Receptor-Mutated Advanced Non-Small Cell Lung Cancer With a Secondary Epidermal Growth Factor Receptor Alteration Whose Disease Had Progressed on First-Line Osimertinib. JCO Precis Oncol. 2025 Jun;9:e2400818. doi: 10.1200/PO-24-00818. Epub 2025 Jun 4. PMID 40466026
- [Derived] Yu HA, Goldberg SB, Le X, Piotrowska Z, Goldman JW, De Langen AJ, Okamoto I, Cho BC, Smith P, Mensi I, Ambrose H, Kraljevic S, Maidment J, Chmielecki J, Li-Sucholeiki X, Doughton G, Patel G, Jewsbury P, Szekeres P, Riess JW. Biomarker-Directed Phase II Platform Study in Patients With EGFR Sensitizing Mutation-Positive Advanced/Metastatic Non-Small Cell Lung Cancer Whose Disease Has Progressed on First-Line Osimertinib Therapy (ORCHARD). Clin Lung Cancer. 2021 Nov;22(6):601-606. doi: 10.1016/j.cllc.2021.06.006. Epub 2021 Jun 25. PMID 34389237
- [Derived] Schmid S, Fruh M, Peters S. Targeting MET in EGFR resistance in non-small-cell lung cancer-ready for daily practice? Lancet Oncol. 2020 Mar;21(3):320-322. doi: 10.1016/S1470-2045(19)30859-9. Epub 2020 Feb 3. No abstract available. PMID 32027845
- See also: ORCHARD study design article. The article includes Module 5 and Module 6 but was written prior to the subsequent modules being added. — http://doi.org/10.1016/j.cllc.2021.06.006